CLINICAL TRIAL: NCT06154655
Title: Hybrid E-zine Health Education Intervention Integrated Within a Mental Health Package for Adolescent Perinatal Depression
Brief Title: Hybrid Health Education Intervention Integrated Within a Mental Health Package for Adolescent Perinatal Depression
Acronym: E-zineMH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ibadan (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Lola Kola, Principal Investigator, University of Ibadan
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: K43TW011046 (NIH)
Record Dates: First submitted 2023-07-13; First posted 2023-12-04 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Perinatal Depression
Keywords: Climate change; Adolescent mental health; Perinatal depression; Health education; Digital health
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Intervention Model Description: A pilot trial will be conducted with 60 perinatal adolescents (30 in the E-zineMH arm and 30 in the control arm). Participants will be assigned to each arms at the beginning of the trial and continue in that arm throughout the trial. Two clinics, with wide geographic seperation will be used in the study. One of the clinics will serve as the intervention clinic and the other will serve as control.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessment will be carried at four months post baseline by 2 outcome assessors blind to study arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): participants will receive health education on climate change included in their routine antenatal care and also have access to the e-magazine accessible through mobile phones
  Interventions: Other: E-zine
- Control Group (No Intervention): participants will receive health education on climate change included in their routine antenatal care

INTERVENTIONS:
Other: E-zine — Health education will be delivered through an electronic magazine
  Arms: Intervention Group

SUMMARY:
The goal of this clinical trial is to develop a hybrid E-zine health education intervention integrated within a mental Health package for adolescent perinatal depression.

The main objective is to:

* Develop a hybrid Health Educational Intervention offering health promotion and disease prevention services on climate change to perinatal adolescents and their caregivers.
* Study the feasibility, acceptability, and usability of E-zineMH in a pilot trial among perinatal adolescents and their caregivers in comparison to a control arm that delivers face-to-face health education in routine antenatal clinics.

Participants will be expected to attend routine antenatal appointments for the duration of the study.

In addition to the face-to-face health education delivered to both groups, the intervention group will be exposed to e-magazines on climate change.

DETAILED DESCRIPTION:
Rising temperatures in tropical regions threaten the mental and overall wellbeing of perinatal adolescents and their infants, increasing their risks of depression and adverse obstetric complications such as miscarriages, preterm birth, low infant birth weight and still births. Integrated health promotion and prevention programmes within collaborative mental health packages in antenatal clinics that recognise the vital roles of family and other caregivers while also offering conveniently accessible services are crucial to implementing behavioural change interventions to address the negative impact of climate change (CCH) in the perinatal adolescent population.

In Nigeria, perinatal adolescents do not enjoy the privileges of division of labour in their households. However, they continue to engage in formal family or informal services (e.g., street hawking, outdoor errands) for extended periods in temperatures of up to 44 °C (111.2 °F). Also, pre-existing multidimensional health vulnerabilities in this population are compounded by (1) continuous exposure to household pollution from indoor cooking fuelled with biomass and use of poisonous pesticides. (2) Droughts and floods from extreme temperatures in tropical climates have increased food insecurity, reduced access to portable clean water, and worsened risks of infectious diseases like malaria and zika virus. The United Nations recommends health education as a key approach to addressing the detrimental effects of CCH. Despite the effectiveness of health education programmes in the antenatal population in areas of nutrition intake, family planning methods, obstetrics complications, and common infections in the perinatal period, very little recognition has been given to themes of CCH as part of essential services in antenatal clinics in primary care in Nigeria. Barriers to implementing environmental health care as part of integrated packages in primary care in Nigeria are high at the needs (context-relevant), service (capacity of providers), and consumer awareness (uptake of services) levels.

Our proposed study addresses context-relevant needs, health workers capacity, and service uptake gaps, by leveraging Virtual space to deliver a Health Education intervention to address impact of CC in perinatal adolescents. Services on health promotion and prevention will be delivered electronically (eHealth) through E-zine (electronic magazine) photos to perinatal adolescents and their caregivers (e.g., parents, partner or guardian). The E-zine would be integrated within an existing hybrid mental health collaborative model in primary care to promote healthy practices to prevent adverse health outcomes of CCH. E-zine photo system development will be guided by key constructs of the Transtheoretical model. Health prevention and promotion content of the E-zine photos will 1) utilise social support to address unhealthy behaviours 2) use context relevant materials to educate and raise awareness on CCH to affect attitudes and beliefs of perinatal adolescents and their caregivers 3) provide risk mitigation information through a pros and cons analysis to create decisional balance, and 4) address self-efficacy to maintain healthy behaviours.

This application builds on the evidence and lessons learned from studies conducted by the PI (Dr. Kola's-K43TW011046-4) in Nigeria on mhGAP -perinatal depression integrated model within primary care, mHealth and technology strategy testing, and implementation system development research. As part of a K43 emerging global leader award, the investigators designed and developed a self-management mobile phone application as an adjunct treatment and part of a hybrid (face-to-face + mobile phone follow-up care) intervention for perinatal adolescents. The intervention was designed to deliver treatment that promote positive mental and overall wellbeing in perinatal adolescents using an age and culturally appropriate approach.

Health Education Intervention in the perinatal population. Health Education Intervention in the perinatal population-HEI have been effective in positively impacting knowledge and behavioural attitudes of pregnant women to enable them control and change their lifestyles for improved health outcomes. Notwithstanding the success of HEI in addressing areas of nutrition intake, family planning methods, obstetrics complications, and common infections of perinatal women in Nigeria, very little recognition have been given to themes of CCH as part of essential services in antenatal clinics in primary care. Barriers to implementing HEI for environmental health care as part of an integrated packages in primary care in Nigeria are high at the needs (context-relevant), service (capacity of providers), and consumer (uptake of services) levels. Specifically, there are no well documented information presenting health needs assessment of CCH in the perinatal adolescents as a way of defining and systematic identifying the unmet needs to this population. Services on health related impact of CCH are currently not part of the health education services delivered in majority of the antennal clinics in Nigeria and care givers also lack knowledge on the relevance of CCH and it impact on the health of perinatal women.

Health decision making for perinatal adolescents. Family members are important and highly influential in the care of pregnant adolescents. Due to the social circumstances surrounding many adolescent pregnancies, and given that many of the girls' pregnancies are unplanned, perinatal adolescents in Nigeria often forfeit the "Power to Decide" on key areas of their living circumstances. Such power are often relinquished to the main care provider who in many cases are their mothers, mothers-in-laws, partners or other family members who are willing to take them on in the period. Their power to make and enact health related decisions are therefore to a large degree influenced by parents, partners or guardians.

Importance of the Knowledge to be Gained Nigerian pregnant adolescents and young mothers encounter significant unmet mental health service needs and significant psychosocial distress, which has contributed to increasing poor mental and public health burden in the country. The proposed study addresses these important service and perinatal adolescent mental health research gaps. Results can be useful for improving our knowledge in implementation research and build sustainable capacity for early prevention and intervention in perinatal adolescent mental health services and sustainable capacity building and supportive supervision models for health care workers in primary health services.

Data Collection:

Methodology for Aim 1: Develop an hybrid Health Educational Intervention of health promotion and disease prevention services on climate change for perinatal adolescents and their caregivers. This will be delivered through E-zine photos and face to face health education, within an existing integrated mental health (E-zineMH) model in primary care. The team will employ a participatory approach that engaging perinatal adolescents, their caregivers, care providers and relevant expert groups to develop new photos and adapt context-relevant ones for E-zine from existing videos of a self-management mobile phone application of a mental care, for perinatal adolescents. E-zinemH will deliver services through photos that are practical, culturally relevant and engaging to the study population and their caregivers.

Step 1. Conduct focus group discussions and one to one key informant interviews with purposively selected health care providers, perinatal adolescents, and care givers of perinatal adolescent groups (n=10 per groups of 3; N=30) to assess current knowledge, attitude and practices of CCH that are injurious to health of perinatal adolescents. Also, the team will explore mitigation plans to identified risks as part of our intervention development plan. Milestone: Context relevant information for the development for E-zineMH Step 2: Expert workshop. A 5 day consultative workshop consisting of 10 maternal and child health specialists, and experts in maternal mental health, environmental health, community health care and digital health will be conducted to develop treatment mitigation plans to identified risks from the activities in step one. The aims of the workshop will be to develop contents for E-zine photos as it relates to CCH and its impact of young mothers; and also to adapt relevant photos of mental and overall wellbeing from existing videos of a self-management application for depression care.

The E-zine structure will be guided by key constructs of the transtheoretical model. For health changes to take place, the transtheoretical model posits the need for 1) social support for changing behaviour, 2) awareness of health benefits and risks as strategies of health promotion and prevention, 3) the need for decisional balance that will be achieved by weighing pros and cons of change, and 4) the need to build self-efficacy -confidence and ability to perform and maintain behaviour to prevent temptation to revert to unhealthy behaviour. These constructs are illustrated in the stages for behavioural changes which include pre-contemplation, contemplation, preparation, action, maintenance.

Blueprint of the E-zineMH system: The investigators anticipate the E-zine system will use positive reinforcement at the end of every theme (session) to encourage the usage of the workshop, system. Praise words with cultural appellations (for example, "Cheers to good health, please proceed to the next session") will be used. Cases of incomplete sessions will also receive encouragement for continuing use (for example "health cannot be bought, just a little bit more effort").

Development of EzineMH prototype.The team will then work with a graphic artist to convert the contents of the narrative scripts into culturally appropriate characters after which will work with the Co-Creation Hub an identified team of local expert programmers with expertise to produce a beta version of the mHealth system (PI, Kola, will lead this effort). The beta version will undergo functional testing through laboratory usability assessments with 3 users (one perinatal adolescent, one caregiver, and one care provider). Based on previous experience it is expected 2 to 3 iterations before testing out in real life in a pilot trial. Milestone: The production of E-zine system to deliver Aim 2: Study the feasibility, acceptability, and usability of e-zineMH in a pilot trial among perinatal adolescents and their caregivers in comparison to a control arm that delivers face to face health education as part of routine health talk in antenatal clinics. A pilot trial will be conducted with 60 randomly selected perinatal adolescents 30 in the E-zineMH arm and 30 in the control arm). The trial is not power to test significance different between study arms but designed to provide enough data on feasibility, acceptability and functionality of the E-zineMH system.

E-zineMH arm: Trained health care providers in primary will deliver health education contents of CCH including effects of extreme weather, heat, flooding, and drought on mental health and overall wellbeing in pregnancy and how adolescent mothers are more at risk due cultural practices. Following the health education session perinatal adolescents present will be invited to participate in the study by a study research assistant who will give details of the study. Next, caregivers of consenting perinatal adolescents will be invited to the clinic the next day after which the care provider and the research assistant will invite them to participate in the study. Perinatal adolescents in the study will receive a mobile phone with password assess to intervention content of E-zineMH. Consenting care givers will be given user names and password to assess of the E-zineMH system online. Trained care providers will follow up perinatal adolescents' use of E-zineMH through separate phone calls to them and their caregivers every two weeks to encourage use.

Control Arm: The treatment package includes health education on CCH: a brief overview of CCH, how it affects pregnant women, how perinatal adolescents are more vulnerable because of cultural norms and practices, impact of CCH on mental (depression and anxiety) and overall wellbeing of perinatal adolescents and their infants, and risk mitigation strategies.

In between baseline assessments and 4 months follow in both intervention and control clinics, health care providers will deliver face to face health education in routine antenatal clinic. A trained senior research assistant with background training in health promotion and prevention will assess health provider's fidelity to delivery of health education with the team developed checklist used during the training.

ELIGIBILITY:
Inclusion Criteria:

Perinatal adolescents aged 16-21 years and below Participants would live in the study area for the 4 months of study participation.

Participants provide informed consent.

Exclusion Criteria:

Patients needing immediate medical attention Patients that would not be available in the neighborhood for up to 4 months duration in the study

Ages: 16 Years to 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Edinburgh Postnatal Depression Scale (EPDS) | Baseline
  The Edinburgh Postnatal Depression Scale (EPDS) is a screening tool for perinatal depression. The cut off for depression is a score equal or greater than 12 point.
Edinburgh Postnatal Depression Scale (EPDS) | Four months after baseline
  The Edinburgh Postnatal Depression Scale (EPDS) is a screening tool for perinatal depression. The cut off for depression is a score equal or greater than 12 point.

SECONDARY OUTCOMES:
WHO Disability Assessment Schedule (WHODAS 2.0) | Baseline
  The WHODAS assesses functioning in psychiatric inpatients. The average scores are comparable to the WHODAS 5-point scale, which allows the clinician to think of the individual's disability in terms of none (0-0.49), mild (0.5-1.49), moderate (1.5-2.49), severe (2.5-3.49), or extreme (3.5-4).
WHO Disability Assessment Schedule (WHODAS 2.0) | Four months after baseline
  The WHODAS assesses functioning in psychiatric inpatients. The average scores are comparable to the WHODAS 5-point scale, which allows the clinician to think of the individual's disability in terms of none (0-0.49), mild (0.5-1.49), moderate (1.5-2.49), severe (2.5-3.49), or extreme (3.5-4).
General Health Questionnaire - 28 (GHQ-28) | Baseline
  General Health Questionnaire - 28 (GHQ-28) questionnaire is used as a screening tool for psychological wellbeing. Participants with scores > 24 may be classified as having psychological disturbances.
General Health Questionnaire - 28 (GHQ-28) | Four months after baseline
  General Health Questionnaire - 28 (GHQ-28) questionnaire is used as a screening tool for psychological wellbeing. Participants with scores > 24 may be classified as having psychological disturbances.

CONTACTS AND LOCATIONS:
Overall Officials: Lola Kola, PhD, Principal Investigator — College of Medicine University of Ibadan
Locations (2):
- Nigeria (2):
  - Abaemu Primary Health Care Center, Ibadan, Oyo State
  - Oranyan Primary Health care centre, Ibadan, Oyo State